CLINICAL TRIAL: NCT00641641
Title: An Open Label Study to Examine the Characteristics of HIV Decay Following Introduction of Combination Antiretroviral Therapy Including Raltegravir During Primary and Chronic HIV Infection
Brief Title: The Effect of Raltegravir on HIV Decay During Primary and Chronic Infection
Acronym: PINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sally Hough, Senior Clinical Project Coordinator, Kirby Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PINT01
Record Dates: First submitted 2008-02-28; First posted 2008-03-24 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: HIV Infection
Keywords: Viral compartments; integrase inhibitor therapy; viral species
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- antiretroviral therapy (Experimental): tenofovir (TDF) + emtricitabine (FTC) as a fixed dose combination administered orally once per day and raltegravir (RAL) administered orally twice per day.
  Interventions: Drug: Tenofovir + emtricitabine + raltegravir.

INTERVENTIONS:
Drug: Tenofovir + emtricitabine + raltegravir. — TDF 300mg once daily + FTC 200mg once daily + RAL 400mg twice daily.
  Other Names: TDF; FTC; RAL

SUMMARY:
The purpose of this study is to measure the decay characteristics of HIV in the blood of patients after taking a combination of anti-HIV drugs, which includes a new class of anti-HIV drug, an integrase inhibitor. This study explores how this new combination of therapy reduces virus in various compartments of the body and immune system.

DETAILED DESCRIPTION:
The study is an open-label study of 3-years duration. This study will be conducted at 4 study sites in Sydney, Australia. Sixteen participants will be recruited comprising 8 participants diagnosed with primary HIV infection (Cohort A) and 8 individuals with chronic HIV infection (Cohort B). All patients must be antiretroviral therapy (ART) naïve and will commence a regimen of combination ART consisting of tenofovir disoproxil fumarate and emtricitabine (TDF/FTC; Truvada) plus the integrase inhibitor, raltegravir. Subjects will be followed for three years with intensive quantification of both plasma RNA and cell associated DNA viral species.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years.
* Provision of written, informed consent.
* Screening plasma HIV RNA > 10,000 copies/mL.
* Screening CD4+ T lymphocyte count > 100 x 10^6)/L.
* No previous antiretroviral therapy.
* Haemoglobin > 115 g/L (female) or > 130 g/L (male).
* Absolute neutrophil count > 1 x 10^9/L.
* Platelet count > 100 x 10^9/L
* Serum bilirubin < 1.5 x ULN.
* Serum alkaline phosphatase < 3 X ULN.
* Serum aspartate aminotransferase (AST) < 3 X ULN.
* Serum alanine aminotransferase (ALT) < 3 X ULN.
* Creatinine clearance > 50mL/min (Creatinine clearance (mL/min) =140 - age x weight creatinine Multiply the result by 1.2 for men).

Cohort A: Primary HIV infection:

Documented acute or early infection diagnosed by:

Acute infection:

< 3 bands on Western Blot and any one of: i. positive p24 antigen ii. positive proviral DNA

Early infection:

i. Positive detuned or BED ELISA result OR ii. Previously negative serology within 6 months of confirmed positive serology.

Cohort B: Chronic HIV infection:

Documented HIV-infection of at least 12 months duration.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Receipt of investigational products within 1 month of study entry.
* Receipt of any of the following within 6 months of study entry:

  * interferon alpha or gamma
  * oral corticosteroids (inhaled or topical corticosteroids are permitted)
  * cyclosporin
  * alkylating agents
  * other immunosuppressive agents
  * rifampin
  * phenytoin
  * phenobarbital
* Documented genotypic (IAS 2007) resistance to tenofovir or emtricitabine from any HIV drug resistance test.
* Any medications contraindicated with Truvada or raltegravir.
* Significant intercurrent illnesses apart from HIV infection such as viral hepatitis (diagnosed by core hepatitis B antigen and/or positive hepatitis B PCR or positive hepatitis C PCR) or any other condition which in the opinion of the investigator would compromise participation in the study.
* History of non-traumatic osteoporotic fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Kelleher, MBBS (Hons) PhD, FRACP, FRCPA, Principal Investigator — Kirby Institute
Locations (4):
- Australia (4):
  - St Vincent's Hospital, Darlinghurst, Sydney, New South Wales
  - 407 Doctors, Sydney, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Taylor Square Private Clinic, Sydney, New South Wales

REFERENCES:
- [Result] Koelsch KK, Boesecke C, McBride K, Gelgor L, Fahey P, Natarajan V, Baker D, Bloch M, Murray JM, Zaunders J, Emery S, Cooper DA, Kelleher AD; PINT study team. Impact of treatment with raltegravir during primary or chronic HIV infection on RNA decay characteristics and the HIV viral reservoir. AIDS. 2011 Nov 13;25(17):2069-78. doi: 10.1097/QAD.0b013e32834b9658. PMID 21860347
- [Result] Murray JM, McBride K, Boesecke C, Bailey M, Amin J, Suzuki K, Baker D, Zaunders JJ, Emery S, Cooper DA, Koelsch KK, Kelleher AD; PINT STUDY TEAM. Integrated HIV DNA accumulates prior to treatment while episomal HIV DNA records ongoing transmission afterwards. AIDS. 2012 Mar 13;26(5):543-50. doi: 10.1097/QAD.0b013e328350fb3c. PMID 22410637
- [Derived] Hey-Cunningham WJ, Murray JM, Natarajan V, Amin J, Moore CL, Emery S, Cooper DA, Zaunders J, Kelleher AD, Koelsch KK; PINT study team. Early antiretroviral therapy with raltegravir generates sustained reductions in HIV reservoirs but not lower T-cell activation levels. AIDS. 2015 May 15;29(8):911-9. doi: 10.1097/QAD.0000000000000625. PMID 25730509
- See also: Peer reviewed publication of trial results — http://www.ncbi.nlm.nih.gov/pubmed/21860347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 5 clinical centres in Sydney
Pre-assignment Details: A screening period of less than 42 days prior to commencement of study drugs was employed
Groups:
- Drug Intervention: Tenofovir+emtricitabine+raltegravir
Period: Overall Study
Arm/Group | Drug Intervention
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Drug Intervention
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Region of Enrollment [Number; unit: participants]
  Australia | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline Plasma HIV RNA (Log Copies/mL)
Description: change was calculated as the mean of 12 assessments minus the baseline value
Time Frame: 12 times within 48 weeks.
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: log copies/mL plasma
Arm/Group | Drug Intervention
Number analyzed (Participants) | 16
log copies/mL plasma | 5.4 (0.6)

ADVERSE EVENTS:
Arm/Group | Drug Intervention
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
Limited cohort (n=16) of exclusively male participants treated with a licensed regimen of combination antiretroviral therapy with the primary focus being a detailed examination of virus decay characteristics

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No